CLINICAL TRIAL: NCT03801668
Title: A Multi-center, Open-label, Randomized Controlled Study of Albumin-bound Paclitaxel Plus S-1 Versus Oxaliplatin Plus S-1 (SOX) as First-line Treatment in Advanced or Recurrent Gastric Adenocarcinoma
Brief Title: Albumin-bound Paclitaxel Plus S-1 Versus SOX as First-line Treatment in Advanced or Recurrent Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Head of the cancer center, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCC008
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Albumin-bound Paclitaxel
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel; S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-P/S-1 (Experimental): Patients in this arm receive chemotherapy with Albumin-bound Paclitaxel plus S-1.
  Interventions: Drug: Albumin-bound Paclitaxel plus S-1
- SOX (Active Comparator): Patients in this arm receive chemotherapy with Oxaliplatin plus S-1.
  Interventions: Drug: Oxaliplatin plus S-1

INTERVENTIONS:
Drug: Albumin-bound Paclitaxel plus S-1 — Albumin-bound Paclitaxel 260mg/m2 IV on D1 plus S-1 80mg/m2 PO (Bid) on D1-14 every 21 days.
  Arms: Nab-P/S-1
Drug: Oxaliplatin plus S-1 — Oxaliplatin 130mg/m2 IV on D1 plus S-1 80mg/m2 PO (Bid) on D1-14 every 21 days.
  Arms: SOX

SUMMARY:
It is a trial to compare the efficacy and safety of Albumin-bound Paclitaxel plus S-1 versus Oxaliplatin plus S-1 (SOX) as first-line treatment in advanced or recurrent gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years;
2. Cytological or histological diagnosis of recurrent or metastatic gastric adenocarcinoma;
3. At least one measurable lesion as defined by RECIST 1.1 criteria;
4. ECOG performance status of 0-1;
5. Estimated life expectancy of at least 3 months;
6. Left ventricular ejection fraction (LVEF) ≥ 50%;
7. Bone marrow function: absolute neutrophil count(ANC) ≥1.5×109 /L, platelet count(PLT) ≥90×109 /L, hemoglobin(HB) ≥90 g/L;
8. Liver and kidney function: Creatinine(Cr)≤1.5 x upper limit of normal range(ULN); alanine glutamate transaminase (ALT) and glutamate transaminase (AST) ≤2.5 x upper limit of normal range (ULN), or ≤5 x upper limit of normal range (ULN)when with hepatic metastases，total bilirubin (TBIL)≤1.5 x upper limit of normal range (ULN), or≤2.5 x upper limit of normal range (ULN) when with Gilbert's syndrome;
9. Not be breast-feeding; men and women of reproductive age are willing to take reliable contraceptive measures during the study;
10. Able and willing to comply with the study plans in this protocol and sign the informed consent;

Exclusion Criteria:

1. Have received chemotherapy before；patients that received neoadjuvant or adjuvant chemotherapy are eligible provided the treatment is completed>6 months prior to first recurrence or metastasis;
2. HER-2 positive;
3. Patients with symptomatic brain metastases;
4. II-IV peripheral neuropathy [NCI-CTCAE 4.03];
5. Anti-HCV antibody positive and HCV-RNA positive; anti-HBV antibody positive with active hepatitis ; anti-HIV antibody positive;
6. Patients with serious systemic infection or other diseases;
7. Allergic to the chemotherapy drugs or the materials in this study;
8. Patients with gastrointestinal bleeding that need clinical intervention;
9. Patients with digestive tract obstruction or oral nutrition difficulty;
10. Have a second malignancy within 5 years prior to registration except for cured carcinoma in situ of cervix uteri, non-melanoma skin cancer;
11. Have participated in other clinical trials within 28 days prior to the first dose of this study;
12. Contraindications to chemotherapy;
13. Patients that researcher consider cannot sign informed consent or complete the study plan due to medical science factor, social factor or psychological reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 3 years
  PFS is defined as time from the start of treatment to progression of disease or death.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | up to 3 years
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
Overall survival (OS) | up to 3 years
  Overall survival is defined as time from the start of treatment until death due to any reason.
Safety as measured by number and grade of adverse events | up to 3 years
  Summary adverse events according to NCI-CTCAE 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Xianglin Yuan, MD,PhD, Study Chair — Tongji Hospital
Locations (1):
- Tongji hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dai YH, Yu XJ, Xu HT, Zhuang L, Zhang MS, Zou YM, Fu Q, Qiu H, Yuan XL. Nab-paclitaxel plus S-1 versus oxaliplatin plus S-1 as first-line treatment in advanced gastric cancer: results of a multicenter, randomized, phase III trial (GAPSO study). Ther Adv Med Oncol. 2022 Aug 12;14:17588359221118020. doi: 10.1177/17588359221118020. eCollection 2022. PMID 35983025